CLINICAL TRIAL: NCT02737774
Title: A Single Armed Phase ⅡStudy of Alternating Icotinib and Chemotherapy for Advanced Non-small Cell Lung Cancer With EGFR Mutation
Brief Title: Alternating Icotinib and Chemotherapy for Advanced Non-small Cell Lung Cancer With EGFR Mutation
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Principal Investigator, Qiming Wang, director, Henan Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HenanCH HX3001
Record Dates: First submitted 2016-04-05; First posted 2016-04-14 (Estimated); Last update posted 2020-07-01 (Actual); Status verified 2020-06

CONDITIONS: Lung Adenocarcinoma
Keywords: Icotinib; chemotherapy; EGFR
MeSH Terms: conditions — Adenocarcinoma of Lung | interventions — icotinib; Pemetrexed; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Icotinib and Pemetrexed/Carboplatin (Experimental): Icotinib: Icotinib for 18 weeks, 125mg Tid，PO. Chemotherapy: pemetrexed 500mg/m2 iv , 4 cycles. carboplatin AUC=5 iv ,4 cycles.
  Then continue with Icotinib, 125mg Tid，PO. until disease progression.
  Interventions: Drug: Icotinib; Drug: Pemetrexed/Carboplatin

INTERVENTIONS:
Drug: Icotinib — All cases that meet the criteria take Icotinib for 18 weeks, If there is no disease progression, then after 14 days of washout period, received 4 cycles of pemetrexed / carboplatin. After the chemotherapy, continue with Icotinib, 125mg Tid，PO. until disease progression.
Drug: Pemetrexed/Carboplatin — All cases that meet the criteria take Icotinib for 18 weeks, If there is no disease progression, then after 14 days of washout period, received 4 cycles of pemetrexed / carboplatin (standard solution, 3 weeks for a cycle of chemotherapy : pemetrexed 500mg/m2 iv , 4 cycles. carboplatin AUC=5 iv ,4 cycles.). After the chemotherapy, continue with Icotinib, 125mg Tid，PO. until disease progression.

SUMMARY:
This is a prospective, open, single-center, phase Ⅱ study to assess the efficacy and safety of alternating Icotinib and chemotherapy for advanced non-small cell lung cancer with EGFR mutation.

ELIGIBILITY:
Inclusion Criteria:

1. Histological or cytological confirmation of non-small cell lung cancer (NSCLC) in phase ⅢB or phase Ⅳ.
2. Positive EGFR mutation(19 exon or 21 exon)。

Exclusion Criteria:

1. Previous usage of EGFR-TKI or antibody to EGFR: gefitinib, erlotinib, herceptin, erbitux.
2. Severe systemic disease out of control such as unstable or uncompensated respiratory,cardiac,liver,renal diseases.
3. Allergic to icotinib
4. metastases of spinal cord, meninges or meningeal.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-04-13 (Actual); Primary Completion 2019-10-25 (Actual); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival | from the day confirmed NSCLC to the day of first detecting progression, up to 24 months

SECONDARY OUTCOMES:
overall survival time | from the day confirmed NSCLC to the day of death, up to 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Qiming Wang, Ph.D, Principal Investigator — Henan Cancer Hospital
Locations (1):
- Henan cancer hospital, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sun X, Zheng Y. Retreatment with icotinib in a patient with metastatic lung adenocarcinoma. Tumori. 2013 May-Jun;99(3):e124-6. doi: 10.1177/030089161309900331. PMID 24158081
- [Background] Zheng Y, Fang W, Deng J, Zhao P, Xu N, Zhou J. Sequential treatment of icotinib after first-line pemetrexed in advanced lung adenocarcinoma with unknown EGFR gene status. J Thorac Dis. 2014 Jul;6(7):958-64. doi: 10.3978/j.issn.2072-1439.2014.07.18. PMID 25093093
- [Background] Wang DS, Patel A, Shukla S, Zhang YK, Wang YJ, Kathawala RJ, Robey RW, Zhang L, Yang DH, Talele TT, Bates SE, Ambudkar SV, Xu RH, Chen ZS. Icotinib antagonizes ABCG2-mediated multidrug resistance, but not the pemetrexed resistance mediated by thymidylate synthase and ABCG2. Oncotarget. 2014 Jun 30;5(12):4529-42. doi: 10.18632/oncotarget.2102. PMID 24980828